CLINICAL TRIAL: NCT07316491
Title: Assessing Possible Improvements to Cosmetic and Functional Outcomes of Penile Split Thickness Skin Grafting With Autologous Fat Graft
Brief Title: Autologous Fat Grafting Beneath Penile Split Thickness Skin Graft Placement During Penile Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Paul Rusilko, Director of Reconstructive Urology, Associate Professor of Urology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY25050015
Record Dates: First submitted 2025-11-26; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Penis/Surgery; Penis/Injuries; Penile Skin; Adult-Acquired Buried Penis
Keywords: Split-Thickness Skin Grafting; Autologous Fat Grafting; Penile Reconstruction
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STSG Alone (Active Comparator): Subjects randomized to this arm of the study will undergo standard-of-care split-thickness skin grafting of their penis without autologous fat grafting. They will undergo the same pre- and post-operative monitoring and complete the same testing as those in the experimental arm of the study.
  Interventions: Procedure: Genitourinary Reconstruction with Split-Thickness Skin Grafting
- STSG with Autologous Fat Grafting (Experimental): Subjects randomized to this arm of the study will undergo standard-of-care split-thickness skin grafting of their penis with autologous fat grafting. For subjects from whom a sufficient quantity of healthy adipose tissue is excised as part of the standard-of-care reconstructive surgery they have elected to undergo, the autologous fat graft will be processed from this specimen and placed between the skin graft and fascia of the penis. For subjects from whom a sufficient quantity of healthy adipose tissue is not excised as part of their standard-of-care reconstructive surgery, lipoaspiration (liposuction) will be performed to harvest fatty tissue that will subsequently undergo minimal processing for grafting.
  Interventions: Procedure: Autologous fat grafting; Procedure: Genitourinary Reconstruction with Split-Thickness Skin Grafting

INTERVENTIONS:
Procedure: Autologous fat grafting — In this intervention, subjects will undergo their standard-of-care reconstructive urologic surgery with penile split-thickness skin grafting as medically indicated for treatment of their underline penile/genitourinary condition(s). In addition to this reconstruction, autologous fat grafting will be performed beneath their penile skin graft. For subjects from whom a sufficient quantity of healthy adipose tissue is excised as part of the standard-of-care reconstructive surgery they have elected to undergo, the autologous fat graft will be processed from this specimen and placed between the skin graft and fascia of the penis. For subjects from whom a sufficient quantity of healthy adipose tissue is not excised as part of their standard-of-care reconstructive surgery, lipoaspiration (liposuction) will be performed to harvest fatty tissue that will subsequently undergo minimal processing for grafting.
  Arms: STSG with Autologous Fat Grafting
Procedure: Genitourinary Reconstruction with Split-Thickness Skin Grafting — Subject eligibility for this study is contingent upon a baseline disease process in which subjects require and are appropriate for genitourinary reconstruction with penile split-thickness skin grafting as their surgical standard of care. Patients in both arms will receive the standard of care reconstruction and split-thickness skin grafting. The donor site for the split-thickness skin graft with be at the discretion of the operating surgeon during the case and will not be affected by enrollment and/or allocation within the trial.

SUMMARY:
The goal of this randomized interventional clinical trial is to learn if placement of a thin layer of fatty tissue (fat graft) beneath a split-thickness skin graft on the surface of the penis improved outcomes of surgery in men who are scheduled to undergo reconstructive surgery on their penis and genitals. This is a randomized study, meaning that half of participants will receive the fat graft with their standard-of-care surgery, and half will have their standard-of-care surgery alone. Fat grafting underneath split-thickness skin grafts in other parts of the body has been shown to improve healing of the skin graft. Both study groups will be followed for specific outcomes through outpatient clinic visits for the first 12 months after their surgery, as well as chart review.

Questions the investigators hope to answer include:

* Does fat grafting improve the pliability and feel of the penile skin after grafting
* Does fat grafting change the penile length after surgery
* Does fat grafting improve sexual function, urinary function, and genital self-image after surgery
* Are there any unforeseen complications related to the fat grafting procedure

Participants will be asked to complete questionnaires related to sexual, urinary, and genital self-image questionnaires before surgery, 3 months after surgery, and 12 months after surgery. Noninvasive testing of the penile skin will also be performed at participants' routine appointments.

DETAILED DESCRIPTION:
The investigators seek to study a novel adipose-based therapeutic strategy to improve cosmetic and function outcomes at the time of penile split-thickness skin graft (STSG) application during penile reconstruction. This entails a therapeutic repurposing of commonly utilized fat and skin grafting protocols to provide a fat-first reconstruction to address each of these limitations in one simple, economical, and widely accessible treatment for point-of-care penile reconstruction. Autologous adipose tissue is ideal as an adjunct to penile split-thickness skin grafting because it: 1) provides immediate, biologic soft tissue coverage with minimal to no donor site burden; 2) remains viable in poorly vascularized wound beds and can be placed as a biologic dressing without specialized microsurgical care; 3) enhances angiogenesis to mitigate risk of infection of deeper structures; 4) mitigates adhesions to underlying structures; and 5) can be used as immediate platform for rapid restoration of cutaneous integrity. By leveraging these techniques, the investigators seek to provide a safe, effective, and available option to augment standard-of-care reconstruction techniques.

Multiple conditions can lead to a need for penile reconstruction. Penile trauma, including burns, penetrating injury, blast injury, and friction injury can irreversibly damage penile skin, leading to a need to resurface the shaft and/or glans of the penis with local tissue flaps or autologous grafts. Infectious processes, most notably Fournier's gangrene, can also lead to loss of penile skin. Finally, adult-acquired buried penis (AABP) disease, a condition wherein the penis becomes trapped by adjacent soft tissues leading to chronic inflammation and loss of penile epithelial integrity, can require surgical excision of penile skin as part of a multicomponent repair. In all of these cases, STSG of the penile shaft is considered standard of care if local flaps, such as scrotal flaps, are not available for reconstruction due to overlapping disease processes. STSGs are commonly utilized to allow for rapid, definitive closure and restoration of the integument.

While STSG graft take on the penis following these processes is successful >95% of the time with restoration of urinary outcomes, patients who have undergone the procedure typically report dissatisfaction with the cosmetic appearance of their penile skin. This is due to adhesion of the STSG to the fixed Buck's deep fascia of the penis, which occurs due to the loss of the mobile Dartos fascia during the time of initial insult/injury. The combination of adhesion and graft contracture/fibrosis can lead to a "plasticky" feeling of the penile skin, which is especially bothersome given the expansile nature of the deep cavernosal bodies during sexual arousal. While current sexual outcomes in patients undergoing penile reconstruction are superior to patients who do not undergo reconstruction, there exists significant room for improvement. There currently exist no off-the-shelf products with proven efficacy in improving outcomes.

Adipose tissue is a prime candidate for this application due to its autologous origin, ease of procurement with minimal-to-no additional donor site morbidity, and abundant availability in patients, alongside its unique reconstructive and regenerative capacities. The use of autologous adipose in delayed tissue reconstruction is well established. However, the full therapeutic potential of adipose tissue remains underexploited. Fat grafting provides immediate soft tissue bulk, enhances angiogenesis, is both immunomodulatory and enhances immunologic homing, and supplies mesenchymal cells for soft tissue healing. Fat grafting is viable in hostile recipient beds including infected/contaminated and poorly vascularized wounds such as the diabetic foot ulcer, irradiated skin, and burn scars.

Grafting of autologous fat tissue is a minimally invasive surgical technique that starts with the harvest of small particles (2-5 mm) of fat tissue from the abdomen or using liposuction. Sometimes, fat graft can be harvested from tissue that is removed for other reasons. This technique utilizes incisions smaller than 5 mm in length and rapid intraoperative processing allowing for immediate transplantation of a patient's own tissue in a single operative procedure. Autologous fat can also be obtained from adipose tissue removed intraoperatively, which is a standard component to AABP repair, and processed intraoperatively for immediate use. This follows a standard fat grafting preparation protocol currently being used for standard of care cases.

A multitude of data exist to support the utility of autologous fat grafting for other disease processes at a variety of anatomic sites. Applications that have been subject to rigorous prior study include:

* Improvement in soft tissue volume, pliability, and skin quality after autologous fat grafting of atrophic amputation stumps
* Improvement in tissue pliability in a porcine burn model
* Improvement in human burn patients when autologous fat grafting was performed beneath a STSG overlying tendon in a burn patient

In the study described herein, participants will undergo the standard-of-care baseline reconstructive surgery for their primary disease process. This will include any necessary debridement, penile degloving, and soft tissue excision of the penis, genitals, and surrounding tissues as indicated by their primary traumatic, infectious, or other disease process. Post-operative wound care will proceed along standard-of-care pathways and will not be altered for the purposes of this protocol.

It is important to recognize that no cell extraction or isolation will be performed in this trial. The fat graft is regulated as a standard surgical procedure with no more than minimal manipulation of the fat tissue. Fat graft injection has been widely adopted by plastic surgeons, dermatologists, and ophthalmologists in clinical practice. Because these are autologous fat grafts that undergo minimal manipulation, they are regulated as a standard surgical procedure and are well-tolerated by patients with minimal safety risks. Only simple processing will be performed with the fat tissue to improve its texture and compliance as is already the standard of care and commonly performed. As autologous fat grafting is well known to soften scarring from trauma, surgical manipulation/incisions, and radiation fibrosis, the investigators believe this approach will be efficacious and well-tolerated due to the common anatomic factors seen in the penis and other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in informed consent
* Loss of penile skin necessitating split-thickness skin grafting for reconstruction
* Willingness to undergo the study interventions and comply with required study procedures
* Is a medical and surgical candidate to undergo standard-of-care split-thickness skin graft reconstruction of the penis after standard preoperative optimization

Exclusion Criteria:

* History of neophallus creation
* A diagnosed disorder of connective tissue or collagen deposition/formation
* The inability to obtain sufficient fat from the surgical specimen or separate lipoharvest donor site to allow the autologous fat tissue processing
* Any medical condition that would preclude safe conduct of the lipoharvest and/or injection procedure per investigator discretion

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Penile Tissue Pliability | 3 and 12 months postoperatively
  The primary outcome of this study will be cutometric assessment of penile tissue pliability following split-thickness skin grafting. This will be measured using established noninvasive, nondestructive techniques that are not expected to cause significant discomfort or distress to patients. The numeric outcome of this, as measured in millimeters, will be directly compared between the experimental and active comparator arms. More pliability is manifested as increased pliability, as measured in millimeters.

SECONDARY OUTCOMES:
Sexual Function | Preoperatively, 3 months postoperatively, and 12 months postoperatively
  Subjects' postoperative sexual satisfaction and sexual function will be assessed using the 15-question validated International Index of Erectile Function questionnaire. Pre- and post-operative total scores (measured on a scale of 0 to 45, where a higher score indicates better sexual satisfaction/function) will be compared in a pairwise manner between arms of the study to determine if autologous fat grafting confers increase improvement on IIEF relative to the active comparator arm.
Urinary Function | Preoperatively, 3 months postoperatively, and 12 months postoperatively
  The Internatonal Prostate Symptom Score (IPSS) validated patient questionnaire will be utilized to assess subjects' satisfaction with their urinary function. This questionnaire includes seven Likert-style questions assessing seven domains of urinary function, where a composite score of 0 represents no symptoms and a composite score of 35 represents maximum symptom burden. The questionnaire also contains one additional quality-of-life question, in which 0 represents maximum aggregate satisfaction with urinary function and 6 represents the worst possible satisfaction with urinary function. The pre- and post-operative scores will be analyzed in a pairwise manner, and the change in scores will be assess between the experimental and active comparator groups.
Genital Self-Image | Preoperatively, 3 months postoperatively, 12 months postoperatively
  Subjects' pre- and post-operative subjective genital self-image will be assessed using the 7-question validated Male Genital Self-Image Scale (MGSIS) questionnaire. Pre- and post-operative total scores (measured on a scale of 7 to 28, where a higher score represents a more positive self-image) will be compared in a pairwise manner between arms of the study to determine if autologous fat grafting confers increase improvement on MGSIS relative to the active comparator arm.
Safety and Surgical Complications | Immediately postoperatively through 12 months, including in-person visits at 7 days, 4 weeks, 3 months, and 12 months postoperatively. A telephone call will also be initiated 6 months postoperatively.
  Patient safety and surgical complications will be closely monitored throughout the convalescence period of the study in the standard manner for their genitourinary reconstruction procedure. Patients will be seen in-person, and contacted via telephone, for assessment of their wounds. At these visits, interval information will be collected to monitor for adverse events, such as graft failure, infection, incisional dehiscence, graft donor site hematoma, and other wound complications. All adverse events will be scored using the Clavien-Dindo classification system, and classified as minor (Clavien-Dindo 1-2) and major (Clavien-Dindo 3-5). The frequency of major and minor complications in the experimental arm will be compared to the frequency in the active comparator arm.
Stretched Penile Length | Intraoperatively, 3 months postoperatively, 12 months postoperatively
  Stretched penile length and associated tissue mobility will be measured and recorded. Average stretched postoperative penile length in the experimental group, as measured in centimeters, will be measured relative to that in the active comparator arm.
Penile Pain and Sensitivity to Monofilament Testing | 3 and 12 months postoperatively
  Penile pain and sensitivity assessment will be performed using standardized protocols for grafting on other areas of the body. These noninvasive methods provide a subjective readout of pain and sensitivity. Specifically, the Semmes Weinstein monofilament test will be used to identify the pressure threshold at which perceptible sensation can be elicited with closed eyes. This is scored on a scale of 1.65-6.65 based on the monofilament sizes within the standard kit. Patients with lower numbers, indicating a smaller monofilament/less pressure can elicit a perceptible response, have greater sensitivity than those with higher numbers. If pain is elicited, they will also be assigned a score on the scale listed above, with a lower score suggestive of lower pain threshold. This will be assessed on the right lateral aspect of the penis, left lateral aspect of the penis, and glans.
Penile Sensitivity to Two-Point Discrimination Testing | 3 and 12 months postoperatively
  The sensitivity of the grafted penile skin will be assessed using the static two-point discrimination test, which is a commonly used test for skin sensitivity testing. In this test, a pair of calipers will be used to determine the spacing at which the patient can detect two discrete points of pressure, as measured in millimeters. A larger distance suggests less sensitivity, while a shorter distance suggests more sensitivity. This will be assessed on the right lateral aspect of the penis, left lateral aspect of the penis, and glans.
Penile Graft Elasticity | 3 and 12 months postoperatively
  Penile graft elasticity will be assessed using noninvasive skin tensiometry. The outcome of this, as measured in mm, will be compared between the experimental and active comparator groups.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Rusilko, DO, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Mercy Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of patients involved in this study, we do not plan on sharing IPD.

REFERENCES:
- [Background] Sivak WN, Ruane EJ, Hausman SJ, Rubin JP, Spiess AM. Decellularized Matrix and Supplemental Fat Grafting Leads to Regeneration following Traumatic Fingertip Amputation. Plast Reconstr Surg Glob Open. 2016 Oct 12;4(10):e1094. doi: 10.1097/GOX.0000000000001094. eCollection 2016 Oct. PMID 27826486
- [Background] Bourne DA, Thomas RD, Bliley J, Haas G, Wyse A, Donnenberg A, Donnenberg VS, Chow I, Cooper R, Coleman S, Marra K, Pasquina PF, Rubin JP. Amputation-Site Soft-Tissue Restoration Using Adipose Stem Cell Therapy. Plast Reconstr Surg. 2018 Nov;142(5):1349-1352. doi: 10.1097/PRS.0000000000004889. PMID 30511990
- [Background] Biyao Z, Gang X, Hai J, Chenwang D, Xuan L. Autologous fat grafting combined with negative pressure wound therapy in severe diabetic foot ulcer: a case study. J Wound Care. 2021 Apr 1;30(Sup4):S38-S40. doi: 10.12968/jowc.2021.30.Sup4.S38. PMID 33856926
- [Background] Piccolo NS, Piccolo MS, Piccolo MT. Fat grafting for treatment of burns, burn scars, and other difficult wounds. Clin Plast Surg. 2015 Apr;42(2):263-83. doi: 10.1016/j.cps.2014.12.009. Epub 2015 Feb 21. PMID 25827568
- [Background] Kenny EM, Egro FM, Ejaz A, Coleman SR, Greenberger JS, Rubin JP. Fat Grafting in Radiation-Induced Soft-Tissue Injury: A Narrative Review of the Clinical Evidence and Implications for Future Studies. Plast Reconstr Surg. 2021 Apr 1;147(4):819-838. doi: 10.1097/PRS.0000000000007705. PMID 33776031
- [Background] Gentile P, Sterodimas A, Calabrese C, Garcovich S. Systematic review: Advances of fat tissue engineering as bioactive scaffold, bioactive material, and source for adipose-derived mesenchymal stem cells in wound and scar treatment. Stem Cell Res Ther. 2021 Jun 2;12(1):318. doi: 10.1186/s13287-021-02397-4. PMID 34078470
- [Background] Dong J, Wu B, Tian W. Adipose tissue-derived small extracellular vesicles modulate macrophages to improve the homing of adipocyte precursors and endothelial cells in adipose tissue regeneration. Front Cell Dev Biol. 2022 Dec 6;10:1075233. doi: 10.3389/fcell.2022.1075233. eCollection 2022. PMID 36561367
- [Background] Theisen KM, Fuller TW, Rusilko P. Surgical Management of Adult-acquired Buried Penis: Impact on Urinary and Sexual Quality of Life Outcomes. Urology. 2018 Jun;116:180-184. doi: 10.1016/j.urology.2018.03.031. Epub 2018 Apr 3. PMID 29625136
- [Background] Seitz AJ, Edalatpour A, Israel JS, Grimes MD, Williams DH, Poore SO. Postoperative Outcomes following Buried Penis Reconstruction: A Single-Institution Experience Using the Wisconsin Classification System. Plast Reconstr Surg. 2024 May 1;153(5):1151-1160. doi: 10.1097/PRS.0000000000010868. Epub 2023 Jun 20. PMID 37337329
- [Background] Staniorski CJ, Myrga JM, Vasan RV, Klein RD, Rusilko PJ. Surgical Outcomes and Prediction of Complications Following High-complexity Buried Penis Reconstruction. J Urol. 2023 Nov;210(5):782-790. doi: 10.1097/JU.0000000000003669. Epub 2023 Aug 16. PMID 37586110
- [Background] Kara O, Teke K, Ciftci S, Ustuner M, Uslubas AK, Bosnali E, Culha MM. Buried penis in adults as a complication of circumcision: Surgical management and long-term outcomes. Andrologia. 2021 Mar;53(2):e13921. doi: 10.1111/and.13921. Epub 2020 Nov 26. PMID 33244793
- [Background] Kumar T, Patel A, Chaffin AE. Use of Suprapubic Panniculus for Split-Thickness Skin Graft in Buried Penis Repair. Eplasty. 2024 Feb 6;24:e6. eCollection 2024. PMID 38476520
- [Background] Flynn KJ, Vanni AJ, Breyer BN, Erickson BA. Adult-Acquired Buried Penis Classification and Surgical Management. Urol Clin North Am. 2022 Aug;49(3):479-493. doi: 10.1016/j.ucl.2022.04.009. Epub 2022 Jun 29. PMID 35931438
- [Background] Falcone M, Preto M, Timpano M, Oderda M, Plamadeala N, Cirigliano L, Blecher G, Peretti F, Ferro I, Gontero P. The outcomes of surgical management options for adult acquired buried penis. Int J Impot Res. 2023 Dec;35(8):712-719. doi: 10.1038/s41443-022-00642-9. Epub 2022 Nov 18. PMID 36400942
- [Background] Thornton SM, Seitz AJ, Edalatpour A, Poore SO. Surgical management of adult acquired buried penis syndrome: A systematic review of patient-reported outcome instruments. J Plast Reconstr Aesthet Surg. 2024 Apr;91:181-190. doi: 10.1016/j.bjps.2024.02.009. Epub 2024 Feb 6. PMID 38422919
- [Background] Deptula P, Fox P. Autologous Fat Grafting in Hand Surgery. J Hand Surg Am. 2021 Jul;46(7):594-600. doi: 10.1016/j.jhsa.2021.02.015. Epub 2021 Apr 13. PMID 33858716
- [Background] Kaur S, Rubin JP, Gusenoff J, Sommers CA, Shamsunder MG, Hume KM, Mehrara BJ. The General Registry of Autologous Fat Transfer: Concept, Design, and Analysis of Fat Grafting Complications. Plast Reconstr Surg. 2022 Jun 1;149(6):1118e-1129e. doi: 10.1097/PRS.0000000000009162. Epub 2022 Apr 11. PMID 35404336